CLINICAL TRIAL: NCT05496712
Title: Effect of Physical Activity in Pregnancy on Maternal and Fetal Human Milk Oligosaccharides: a Pilot Study
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 26-380 ex 13/14
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy, Physical Activity
Keywords: Human Milk Oligosaccharides
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — maternal venous blood (serum / plasma); cord blood (serum / plasma); placenta tissue (RNA later, cryo specimen); maternal urine; maternal saliva; vaginal swabs;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study investigates the interaction of maternal physical activity (PA) and body composition during pregnancy with prenatal Human Milk Oligosaccharide (HMO) concentrations, and assesses associations of HMOs with fetal/neonatal outcomes.

DETAILED DESCRIPTION:
Maternal obesity is a known risk factor for adverse short- and long-term health outcomes for the offspring. In non-pregnant individuals, obesity can alter glucose and fat metabolism, and induce a low-grade inflammation. Pregnancy is a natural state of low-grade inflammation in the mother and the feto-placental unit, and the severity of this inflammation increases with higher pre-gravid BMI. Consequently, in pregnant women, obesity could account for an altered intrauterine environment that might affect fetal development and programming.

Regular physical activity (PA) is associated with a reduced inflammatory state. PA has been determined as a major factor contributing to fetal growth and body composition, besides maternal nutrition, gestational diabetes and obesity.

Human milk oligosaccharides (HMOs), highly bioactive factors in breast milk, but also present in the systemic circulation of pregnant women, may be one of the factors altered by metabolic changes seen in obesity, which might have an impact on the health of the offspring. HMOs have been implicated in multiple beneficial effects for the breast-fed infant, and also have anti-inflammatory and immuno-modulating effects.

HMOs are found in the urine of pregnant and lactating women, indicating that HMO circulate in the maternal blood system during pregnancy and throughout lactation. HMOs can also be detected in umbilical cord blood, suggesting either transplacental transfer or fetal production and release, raising the question whether maternal and fetal HMOs have a health impact on mother and fetus and, consequently, could be monitored as potential biomarkers for adverse pregnancy outcomes.

More than 150 HMO structures are known, and HMO composition and concentration in breast milk vary significantly between mothers and also within one mother due to different stages of lactation. Genetic factors and potentially also environmental factors contribute to the composition of HMOs in an individual. Different prenatal HMO profiles could potentially affect maternal and fetal health. Whether HMO composition and concentrations are different in women with overweight or obesity is not known. Exposure to a changed intrauterine environment could potentially pose a risk factor for certain pregnancy outcomes or cause aberrant fetal programming. At the same time, lifestyle factors that can counteract some obesity-induced metabolic changes such as physical activity and diet could potentially also have an effect on HMO concentration/composition.

The overall objective of the study is to investigate the interaction of maternal physical activity on HMOs in maternal and fetal circulation.

Specific Aims are:

* To longitudinally determine maternal HMO concentration and composition during gestation to describe variability and temporal changes.
* To assess fetal HMO concentration and composition to gain insight about origin: comparison arterial vs. venous cord blood; maternal vs. fetal HMOs.
* To investigate associations of maternal and fetal HMOs with maternal body mass index/physical activity, and fetal growth/body composition.

ELIGIBILITY:
Inclusion Criteria:

* ongoing pregnancy no later than 14 weeks of gestation
* giving informed consent

Exclusion Criteria:

* not wanting to give birth at the university hospital
* gestational age > 14th week of gestation
* multiple pregnancy
* 3 or more consecutive miscarriages
* increased risk ≥ 1:100 after combined test (minimum parameters: maternal age, Fetal CRL, nuchal translucency, nasal bone and maternal biochemistry - free-ß-hCG and PAPP-A) and no NIPT (Non-Invasive Prenatal Testing) or no invasive testing for chromosomal anomalies
* fetal anomalies which are associated with possible growth or genetic anomalies
* smoking
* pre-pregnancy diabetes type 1 or 2 (T1D, T2D)
* maternal metabolic risk factors (autoimmune conditions, increased risk for thromboembolic events needing anticoagulative therapy)
* pre-pregnancy hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible are women with an on-going healthy pregnancy. Physical activity will be objectively measured by accelerometer. Women will be recruited as soon as possible in their pregnancy, but not after the 14th week of gestation. They will be recruited through the outpatient clinic at the Department of Obstetrics, Medical University Graz.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Human milk oligosaccharides (HMO) composition and concentration in maternal blood | 6 months
  HMOs will be analysed in maternal blood by high pressure liquid chromatography (HPLC) with fluorescence detection
Human milk oligosaccharides (HMO) composition and concentration in fetal blood | 6 months
  HMOs will be analysed in fetal (umbilical cord) blood by high pressure liquid chromatography (HPLC) with fluorescence detection
Human milk oligosaccharides (HMO) composition and concentration in maternal urine | 6 months
  HMOs will be analysed in maternal urine by high pressure liquid chromatography (HPLC) with fluorescence detection
Human milk oligosaccharides (HMO) composition and concentration in colostrum | 6 months
  HMOs will be analysed in colostrum by high pressure liquid chromatography (HPLC) with fluorescence detection

SECONDARY OUTCOMES:
Fetal growth | 6 months
  fetal growth (longitudinal ultrasound measurements)
Birth weight | 6 months
  infant weight at birth (scale)
Fetal body fat mass | 6 months
  Fetal body fat mass (measured by air displacement plethysmography, PEAPOD)
Fetal fat free mass | 6 months
  Fat free mass (measured by air displacement plethysmography, PEAPOD)
Subcutaneous adipose tissue thickness | 6 months
  Subcutaneous adipose tissue thickness (measured by lipometer at 15 defined body sites)
Cord blood metabolic parameters - Glucose | 6 months
  Glucose
Cord blood metabolic parameters- Insulin | 6 months
  Insulin
Cord blood metabolic parameters - C-Peptide | 6 months
  C-peptide
Cord blood metabolic parameters - erythropoietin | 6 months
  Erythropoietin (measure for fetal hypoxia)
Cord blood metabolic parameters - lipid profile | 6 months
  lipid profile (triglycerides, phospholipids, free fatty acids, HDL proteome)
Cord blood metabolic parameters - Cytokines | 6 months
  Cytokines
Maternal body composition - BMI | 6 months
  Body mass index (BMI)
Maternal body composition - weight gain | 6 months
  gestational weight gain
Maternal body composition - subcutaneous adipose tissue thickness | 6 months
  subcutaneous adipose tissue thickness (measured by lipometer at 15 defined body sites)
Maternal parameters - Glucose | 6 months
  glucose
Maternal parameters - Insulin | 6 months
  insulin
Maternal parameters - C-Peptide | 6 months
  C-peptide
Maternal parameters - Leptin | 6 months
  Leptin
Maternal parameters - Adiponectin | 6 months
  Adiponectin
Maternal parameters - Liquid profile | 6 months
  Lipid profile (triglycerides, phospholipids, free fatty acids, HDL/LDL/total cholesterol)
Maternal parameters - Cytokines | 6 months
  Cytokines
Placental outcomes - Utero-placental blood flow | 6 months
  Utero-placental blood flow (ultrasound/Doppler)
Placental outcomes - fetal-placental blood flow | 6 months
  fetal-placental blood flow (ultrasound/Doppler)
Placental volume | 6 months
  placental volume (ultrasound)
Placental outcomes - Cytokine mRNA | 6 months
  Cytokine mRNA
Placental outcomes - Macrophage density | 6 months
  Macrophage density (number/tissue protein)
Placental outcomes - TREG density | 6 months
  Treg density (number/tissue protein)
Placental outcomes - placental volume | 6 months
  placental volume
Placental outcomes- transcriptomic profile | 6 months
  Transcriptomic profile, RNAseq on a NovaSeq 6000 (Illumina)
Placental outcomes - epigenomic profile | 6 months
  Epigenomic profile measured by DNA methylation
Vaginal Microbiome | 6 months
  From the extracted DNA, 16S rRNA genes will be amplified using specific primers for bacterial and archaeal communities. The amplicons obtained will be prepared for Illumina MiSeq Sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Bence Csapo, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

REFERENCES:
- [Derived] Garcia MG, Hamann E, Huhn EA, Forbes K, Roser P, Weiser-Fuchs MT, Dieberger AM, Csapo B, Obermayer-Pietsch B, Poppel MNMV, Fluhr H, Jantscher-Krenn E, Blois SM. Maternal Galectins and Glucose Regulation in Pregnancy: Chronic vs. Acute Metabolic Adaptations. Diabetes Metab J. 2025 Dec 29. doi: 10.4093/dmj.2025.0401. Online ahead of print. PMID 41299831